CLINICAL TRIAL: NCT01181557
Title: Prospective Evaluation of Quality of Life in Patient With Rectal Cancer
Brief Title: A Questionnaire to Assess the Quality of Life of Rectal Cancer Patients With or Without Stoma
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Alberto Vannelli, Ermanno Leo, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Other Study IDs: INT-D176768
Record Dates: First submitted 2010-04-01; First posted 2010-08-13 (Estimated); Last update posted 2010-08-13 (Estimated); Status verified 2008-07

CONDITIONS: Rectal Cancer
Keywords: quality of life
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- rectal cancer with stoma: rectal cancer submitted to rectal anterior resection with stomia (RARS). Differences in QoL between the two groups were analyzed during three time: first preoperative, second postoperative and latter six month after stoma reconversion
- rectal cancer without stoma: rectal cancer submitted to rectal anterior resection (RAR) Differences in QoL between the two groups were analyzed during three time: first preoperative, second postoperative and latter six month later
- anterior resection of rectum: patients with rectal cancer submitted to RAR and patients with rectal cancer submitted to RARS

SUMMARY:
The aim of the present prospective study was to evaluate the prediction accuracy of EORTC QLQ-C30/C38 questionnaire in rectal cancer patient(RC). This study was designed to investigate how the quality of life (QoL) of patients with rectal cancer changes with time after cancer or after stomia.

Eligible subjects were consecutively enrolled in the investigators' Institute and subjected to EORTC QLQ-C30/C38 questionnaire.

DETAILED DESCRIPTION:
Eligibility criteria: Italian people with adenocarcinoma of rectum. Exclusion criteria consisted of age younger than 18 years, history of psychiatric illness, and preoperative radiotherapy.

Outcome measures: patient was carried out using a EORTC QLQ-C30/C38 questionnaire.To determine how surgery affects QoL, we divided patients into two groups: first rectal cancer submitted to rectal anterior resection(RAR) and latter rectal cancer submitted to rectal anterior resection with stomia(RARS). Differences in QoL between the two groups were analyzed during three time: first preoperative, second postoperative and latter six month later of after the stoma reconversion in RARS patients

ELIGIBILITY:
Inclusion Criteria:

* Rectal cancer

Exclusion Criteria:

* Age younger than 18 years
* History of psychiatric illness
* Preoperative radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients admitted to hospital for rectal cancer, Italian resident older than 18 years, without history of psychiatric illness, or preoperative radiotherapy, dived in two cohorts patient with stoma after surgery and patients without stoma after surgery
Sampling Method: Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2008-09; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Questionnaire number 1, to Assess the Quality of Life of Rectal Cancer Patients With or Without Stoma | three month: first admission in hospital preoperative time
  Two cohort in preoperative time: first EORTC QLQ-C30/C38 questionnaire in rectal cancer submitted to RAR and latter in rectal cancer submitted to RARS.

SECONDARY OUTCOMES:
Questionnaire number 2, to Assess the Quality of Life of Rectal Cancer Patients With or Without Stoma | Three months postoperative time
  Two cohort in postoperative time (three months after surgical procedure): first EORTC QLQ-C30/C38 questionnaire in rectal cancer submitted to RAR and latter in rectal cancer submitted to RARS.
Questionnaire number 3, to Assess the Quality of Life of Rectal Cancer Patients With or Without Stoma | Six months after postoperative time
  Two cohort in postoperative time (six months after postoperative time): first EORTC QLQ-C30/C38 questionnaire in rectal cancer submitted to RAR and latter in rectal cancer submitted to RARS.

CONTACTS AND LOCATIONS:
Overall Officials: alberto vannelli, MD, Study Director — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milano, Milan, Italy, Italy